CLINICAL TRIAL: NCT02007408
Title: Comparison of Lidocaine Spray and Paracervical Block Application for Pain Relief During First-trimester Surgical Abortion: a Randomized, Double-blind, Placebo-controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gökhan Açmaz, MD, Kayseri Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KERH
Record Dates: First submitted 2013-11-25; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Pain Score
Keywords: abortion; analgesia; paracervical block; lidocaine spray
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Obstetrical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo group (Placebo Comparator)
- Paracervical block plus lidocaine spray (Active Comparator): Lidocaine injection+Lidocaine spray received PCB with 2 ampoules of lidocaine solution plus 2 pumps (20 mg=2 pumps) of 10% lidocaine spray
  Interventions: Drug: Paracervical block + lidocaine spray
- paracervical block plus isotonic saline spray (Active Comparator): 2 ampoules of lidocaine solution (20 mg Lidocaine HCl+0.0125 mg epinephrine/ml) plus isotonic spray
  Interventions: Drug: Paracervical block
- only lidocaine spray (Active Comparator): paracervical block with saline solution plus 10% lidocaine spray
  Interventions: Drug: Lidocaine spray

INTERVENTIONS:
Drug: Paracervical block
  Arms: paracervical block plus isotonic saline spray
Drug: Lidocaine spray
  Arms: only lidocaine spray
Drug: Paracervical block + lidocaine spray
  Arms: Paracervical block plus lidocaine spray

SUMMARY:
Objective: The investigators sought to investigate the analgesic efficiency of lidocaine spray, paracervical block (PCB) with lidocaine and PCB with lidocaine plus lidocaine spray combination in patients undergoing first-trimester surgical abortion.

Methods: A randomized, double-blind, placebo-controlled clinical trial was conducted on 108 women with the request of pregnancy termination.The subjects were randomly assigned into four groups: PCB (n=27), lidocaine spray (n=27), PCB plus lidocaine spray (n=27) and placebo(n=27).Intraoperative and postoperative pain scores were measured with a standard Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

Age >18 years Single Pregnancy <7 weeks of gestation

Exclusion Criteria:

Incomplete abortion Early pregnancy failure Acute cervicitis Untreated pelvic inflammatory disease Cervical stenosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Gökhan Açmaz, Kayseri, Turkey (Türkiye)